CLINICAL TRIAL: NCT00627757
Title: Changes in Enteroendocrine and Neuroendocrine Axes in Patients With Weight Gain After Treatment With Antipsychotics
Brief Title: Antipsychotic Medicine and Metabolic Syndrome
Acronym: AMMS1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Henrik Lublin MD DMSc, Chairman and Associate Pofessor of Psychiatry, Psychiatric University Center Glostrup Copenhagen University Hospitals
Other Study IDs: HC-2007-0069; 2602-706
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; weight gain; antipsychotic drugs; Metabolic syndrome and treatment with antipsychotic drugs
MeSH Terms: conditions — Metabolic Syndrome; Weight Gain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Food challenge test: Patients
  51 patients included
- C: Controls 93 healthy controls are included

SUMMARY:
The purpose of the study is to determine whether antipsychotic treatment is influence psychiatric patients due to endocrine and metabolic status and a quality of life.

The investigators expect, that 30-50% of patients will show pharmacon - gene induced weight gain (> 7% of initial bodyweight) while the rest of patients will maintain unaltered bodyweight.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate status of neuro-and enteroendocrine axes with focus on beta - cell function in relation to insulin resistance, lipid profile abnormalities and inflammations adipokins in patients during treatment with antipsychotics (AP) in relation to weight gain.

The second aim is to evaluate the connection between weight gain and patients´ own perception of their quality of life and health.

ELIGIBILITY:
Inclusion Criteria:

* gender : male
* age: 18-45
* treatment with minimum one Antipsychotic drug (AP)
* ethnicity: caucasians
* consent given to take part in the project

Exclusion Criteria:

One criteria is sufficient to exclude patients from the study:

* compliance problems
* unable to read, write and talk Danish
* patients with major lung-,heart-, lever- and kidney problems
* patients with diagnose and treatment for Diabetes 1 and 2
* patients taking cholesterol-reducing, weight-reducing and antihypertensive medication
* patients with abuse of alcohol or drugs
* patients who are under duress §
* patients who have been mentally ill for more than 15 years
* patients with diagnosis/treatment for NIDDM/IDDM

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 patients and 100 control persons. Patients should be treated with minimum one antipsychotic drug and hospitalized or treated as out-patients at Glostrup, Ballerup or Gentofte hospitals.
  Controls will be chosen from the database at Institute of Health and Prevention, Glostrup.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Lublin, MD DMSc, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Psychiatric University Center Glostrup, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Ebdrup BH, Knop FK, Madsen A, Mortensen HB, Sogaard B, Holst JJ, Szecsi PB, Lublin H. Glucometabolic hormones and cardiovascular risk markers in antipsychotic-treated patients. J Clin Psychiatry. 2014 Sep;75(9):e899-905. doi: 10.4088/JCP.13m08820. PMID 25295432